CLINICAL TRIAL: NCT02912221
Title: Influence of Increased Physical Activity on Patient Reported Measures of Disease Activity in Inflammatory Arthritis
Brief Title: Stepping Up For Inflammatory Arthritis
Acronym: SUFIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 825214
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Arthritis, Psoriatic; Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will be reimbursed for participation in the study but will not receive other encouragements for meeting fitbit and step count goals
- Incentive (Active Comparator): An incentive will be used for this arm to encourage participants to meet their step goals
  Interventions: Other: Incentive

INTERVENTIONS:
Other: Incentive — Both groups will receive fitbits to track their physical activity, however one arm of the study may receive additional incentives to achieve their step count goal.
  Arms: Incentive

SUMMARY:
This study will examine the benefits of a monitored physical activity program for participants with rheumatoid arthritis (RA) or psoriatic arthritis (PsA) using a wearable activity device (e.g.fitbit). The goals of this pilot study are to examine 1) whether an incentive is better than no incentive in maintaining an increased level of physical activity and 2) the benefits of physical activity on patient reported disease activity in inflammatory arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) and psoriatic arthritis (PsA) are chronic, systemic inflammatory disorders affecting 1-2% of the US population. Ongoing chronic inflammation and lack of exercise due to arthritis are each associated with pain, fatigue, depression, muscle loss, obesity, and development of chronic diseases such as cardiovascular disease and diabetes, all of which impact physical functioning and quality of life. Increases in physical activity can significantly impact each one of these outcomes and are likely to positively impact a patients experience of their disease. This study will examine the benefits of a monitored physical activity program. This study will use a wearable activity device (e.g. fitbit) to monitor step counts and will incentivize one group to achieve higher step counts than the control group. The primary goal of this pilot study will be to determine whether one incentive (loss aversion) is better than no incentive in increasing step counts and maintaining an increased level of physical activity.

Additional outcomes of interest are patient reported disease activity (using the RAPID3 patient reported outcome) and physician measured disease activity, quality of life assessments and weight loss.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of RA or PsA by a rheumatologist
* Followed by a Penn rheumatologist
* Age 18-80
* A RAPID3 score of 3
* An active email account
* Owns a smart phone and able to download an application
* Willing to take internet based surveys weekly and allow data from a smart phone application to be uploaded

Exclusion Criteria:

* Inability to walk or regular use of a wheel chair or assistive device (e.g., walker or cane)
* Hospitalization within the past 30 days
* Heart or lung disease that precludes participation in an exercise study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-11-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Days Goal Met | 12 Weeks
  The primary outcome will be percent of days meeting goal during the intervention period

SECONDARY OUTCOMES:
RAPID3 | 26 Weeks
  Comparison of RAPID3 score and amount of physical activity
Psoriasis | 26 Weeks
  Physician-assessed psoriasis severity as measured by body surface area (BSA) involved in patients with concurrent psoriasis.
Patient Feedback | 14 Weeks and 26 Weeks
  Patient feedback as determined by qualitative surveys taken at Week 14 and Week 26
Sleep Disturbance and Fatigue | 26 Weeks
  Changes in sleep disturbance and fatigue as determined by PROMIS forms.
Completion of Activities by Study Participants (Feasibility) | 26 Weeks
  Percentage completion of study activities (weekly questionnaires and transmission of activity into Epic

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Ogdie-Beatty, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital at the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share the results of the study after completion of the study through publication in a peer-reviewed journal. Investigators wishing to use the de-identified dataset for additional analyses can contact the PI after publication.